CLINICAL TRIAL: NCT06596239
Title: Hard- and Soft-tissue Changes Following Class III Treatment With the Lower-Clear-Plate-Based Intermaxillary Traction Versus the Removable Mandibular Retractor: a Two-arm Randomized Controlled Clinical Trial
Brief Title: Evaluating the Effectiveness of the Lower-Clear-Plate-Based Intermaxillary Traction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-4-2024
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Class III Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lower-clear-plate-based intermaxillary traction (LCP-IMT) (Experimental): Patients in this group will be treated using the LCP-IMT technique.
  Interventions: Device: lower-clear-plate-based intermaxillary traction (LCP-IMT)
- Removable mandibular retractor (RMR) (Active Comparator): Patients in this group will be treated using the RMR appliance.
  Interventions: Device: Removable mandibular retractor (RMR)

INTERVENTIONS:
Device: lower-clear-plate-based intermaxillary traction (LCP-IMT) — The patient is instructed to apply elastics between the upper molar bands and the hooks on the lower clear plates.
  Arms: Lower-clear-plate-based intermaxillary traction (LCP-IMT)
Device: Removable mandibular retractor (RMR) — An appliance is worn on the upper jaw, which affects the lower jaw by using an inferiorly extended labial bow.
  Arms: Removable mandibular retractor (RMR)

SUMMARY:
Patients at the Orthodontic Department of the University of Damascus Dental School will be examined, and subjects who meet the inclusion criteria will be included. Then, initial diagnostic records (diagnostic gypsum models, internal and external oral photographs, and radiographic images) will be studied to ensure the selection criteria are accurately matched.

This study compares two groups of patients with mild to moderate skeletal Class III in the late mixed occlusion stage. Experimental group: the patients in this group will be treated with Lower-Clear-Plate Based Intermaxillary Traction Control group: the patients in this group will be treated using the Removable Mandibular Retractor (RMR).

DETAILED DESCRIPTION:
There are different methods of correcting Class III deformity in Orthodontics. Lower-clear-plate-based intermaxillary traction has been shown to be an effective method of managing these cases. This treatment modality has not been compared with the well-known appliance (the removable mandibular retractor; RMR). Therefore, the current study compares both groups of growing children with Class III malocclusion. The study design is a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Class III dental malocclusion at the molar relationship, according to Angle's classification
* Presence of an anterior crossbite on two or more teeth or an edge-to-edge relationship at the anterior teeth
* Mild to moderate skeletal Class III in the late mixed occlusion stage (9-13 years old) or the beginning of permanent occlusion (not exceeding 13 years old; ANB = +1 to -4 degrees)
* Normal or horizontal growth pattern (MM ≤ 35; SN.ManP ≤ 40)
* Normal or labial inclination of the lower incisors (IMPA = 85 to 100 degrees)
* Patient's willingness to cooperate during the orthodontic treatment period

Exclusion Criteria:

* Class III skeletal relationship caused solely by the maxillary recession (SNA < 78 and a normal SNB angle)
* An indication of RME
* Presence of clear asymmetry (deviation of mandibular midline more than 2 mm from facial midline)
* Presence of any craniofacial syndromes (such as cleft lip or palate)
* Systemic diseases; previous facial trauma; and Previous orthodontic treatment.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Change in the SNA angle | Time 1: one day before the start of treatment; Time 2: one day after the end of active treatment which is expected to occur within three months in the LCP-IMT group and five months in the RMR group
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the position of the upper jaw in the cephalometric analysis in the anteroposterior direction.
Change in the SNB angle | Time 1: one day before the start of treatment; Time 2: one day after the end of active treatment which is expected to occur within three months in the LCP-IMT group and five months in the RMR group
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the position of the lower jaw in the cephalometric analysis in the anteroposterior direction.
Change in the ANB angle | Time 1: one day before the start of treatment; Time 2: one day after the end of active treatment which is expected to occur within three months in the LCP-IMT group and five months in the RMR group
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the spatial relationship between the upper and lower jaws in the cephalometric analysis in the anteroposterior direction.
Change in the S.N.Pog angle | Time 1: one day before the start of treatment; Time 2: one day after the end of active treatment which is expected to occur within three months in the LCP-IMT group and five months in the RMR group
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the position of the chin in the cephalometric analysis in the anteroposterior direction.
Change in the SN-MaxP angle | Time 1: one day before the start of treatment; Time 2: one day after the end of active treatment which is expected to occur within three months in the LCP-IMT group and five months in the RMR group
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the relationship between the upper jaw plane and the cranial base in the vertical direction of cephalometric analysis.
Change in the SN-ManP angle | Time 1: one day before the start of treatment; Time 2: one day after the end of active treatment which is expected to occur within three months in the LCP-IMT group and five months in the RMR group
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the relationship between the lower jaw plane and the cranial base in the vertical direction of cephalometric analysis.
Change in the MaxP.ManP angle | Time 1: one day before the start of treatment; Time 2: one day after the end of active treatment which is expected to occur within three months in the LCP-IMT group and five months in the RMR group
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the amount of vertical divergence between the upper and lower jaws in the cephalometric analysis.
Change in the Bjork sum (NS-Ar + S-Ar-Go +Ar-Go-Me) | Time 1: one day before the start of treatment; Time 2: one day after the end of active treatment which is expected to occur within three months in the LCP-IMT group and five months in the RMR group
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees.
Change in the Wits appraisal | Time 1: one day before the start of treatment; Time 2: one day after the end of active treatment which is expected to occur within three months in the LCP-IMT group and five months in the RMR group
  Lateral cephalometric images were taken for each patient. This was measured millimetres horizontally from the projection of points A (AO) and B (BO) along the functional occlusal plane.
Change in the U1.SN angle | Time 1: one day before the start of treatment; Time 2: one day after the end of active treatment which is expected to occur within three months in the LCP-IMT group and five months in the RMR group
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the relationship between the upper central incisor axis and the cranial base in the anteroposterior direction of cephalometric analysis.
Change in the L1-GoMe angle | Time 1: one day before the start of treatment; Time 2: one day after the end of active treatment which is expected to occur within three months in the LCP-IMT group and five months in the RMR group
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the relationship between the lower central incisor axis and the mandibular plane in the anteroposterior direction of cephalometric analysis.
Change in the overbite (Ovb) | Time 1: one day before the start of treatment; Time 2: one day after the end of active treatment which is expected to occur within three months in the LCP-IMT group and five months in the RMR group
  Lateral cephalometric images were taken for each patient. This was measured in millimetres vertically from the upper to the lower central incisors.
Change in the overjet (Ovj) | Time 1: one day before the start of treatment; Time 2: one day after the end of active treatment which is expected to occur within three months in the LCP-IMT group and five months in the RMR group
  Lateral cephalometric images were taken for each patient. This was measured millimetres Horizontally from the upper to the lower central incisors.

SECONDARY OUTCOMES:
Change in the Soft tissue convexity angle | Time 1: one day before the start of treatment; Time 2: one day after the end of active treatment which is expected to occur within three months in the LCP-IMT group and five months in the RMR group
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle is to evaluate the profile of the face. It is formed by the intersection of two lines: one from the glabella (the area between the eyebrows) to the subnasale (the point where the nose meets the upper lip), and another from the subnasale to the pogonion (the most forward point on the chin in the cephalometric analysis in the anteroposterior direction.
Change in the Ls-Esth measurement | Time 1: one day before the start of treatment; Time 2: one day after the end of active treatment which is expected to occur within three months in the LCP-IMT group and five months in the RMR group
  Lateral cephalometric images were taken for each patient. This was measured in millimetres from the Labrale superius and E-Line of Ricketts.
Change in the Li-Esth measurement | Time 1: one day before the start of treatment; Time 2: one day after the end of active treatment which is expected to occur within three months in the LCP-IMT group and five months in the RMR group
  Lateral cephalometric images were taken for each patient. This was measured in millimetres from the Labrale inferius and E-Line of Ricketts.
Change in the Nasolabial angle | Time 1: one day before the start of treatment; Time 2: one day after the end of active treatment which is expected to occur within three months in the LCP-IMT group and five months in the RMR group
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the relationship between the nose and the upper lip in the cephalometric analysis in the anteroposterior direction.
Change in the Mento-labial angle | Time 1: one day before the start of treatment; Time 2: one day after the end of active treatment which is expected to occur within three months in the LCP-IMT group and five months in the RMR group
  Lateral cephalometric images were taken for each patient, and this angle was measured in degrees. This angle represents the relationship between the chin and the lower lip in the cephalometric analysis in the anteroposterior direction.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Younis Hajeer, Study Chair — Yes
Locations (1):
- Department of Orthodontics, Faculty of Dentistry, University of Damsacus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Husson AH, Burhan AS, Hajeer MY, Nawaya FR. Evaluation of the dimensional changes in the mandible, condyles, and the temporomandibular joint following skeletal class III treatment with chin cup and bonded maxillary bite block using low-dose computed tomography: A single-center, randomized controlled trial. F1000Res. 2023 Mar 13;12:264. doi: 10.12688/f1000research.130941.1. eCollection 2023. PMID 37008891
- [Background] Garattini G, Levrini L, Crozzoli P, Levrini A. Skeletal and dental modifications produced by the Bionator III appliance. Am J Orthod Dentofacial Orthop. 1998 Jul;114(1):40-4. doi: 10.1016/s0889-5406(98)70235-5. PMID 9674678
- [Background] Saleh M, Hajeer MY, Al-Jundi A. Short-term soft- and hard-tissue changes following Class III treatment using a removable mandibular retractor: a randomized controlled trial. Orthod Craniofac Res. 2013 May;16(2):75-86. doi: 10.1111/ocr.12007. Epub 2012 Nov 8. PMID 23323964
- [Background] Majanni AM, Hajeer MY. The Removable Mandibular Retractor vs the Bone-anchored Intermaxillary Traction in the Correction of skeletal class III Malocclusion in children: A Randomized Controlled Trial. J Contemp Dent Pract. 2016 May 1;17(5):361-71. doi: 10.5005/jp-journals-10024-1856. PMID 27443361
- [Background] Baccetti T, Tollaro I. A retrospective comparison of functional appliance treatment of Class III malocclusions in the deciduous and mixed dentitions. Eur J Orthod. 1998 Jun;20(3):309-17. doi: 10.1093/ejo/20.3.309. PMID 9699409